CLINICAL TRIAL: NCT05016622
Title: Safety and Efficacy of Booster Doses of COVID-19 Vaccine in Immunocompromised Patients With a Cancer Diagnosis
Brief Title: Booster Dose Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to decreased level of engagement and available funding, PI determined it appropriate to close the study prior to visit occurring. IRB approved.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other); National Cancer Institute (NCI) (NIH); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021-13204; 2UG1CA189859-06 (NIH); IRV-BC0004-22 (Other Grant/Funding Number: Leukemia & Lymphoma Society); 3P30CA013330-49S3 (NIH)
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Cancer
Keywords: COVID-19; Booster
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Booster dose (Experimental)
  Interventions: Biological: BNT162b2 vaccine

INTERVENTIONS:
Biological: BNT162b2 vaccine — Administer an additional dose of the BNT162b2 mRNA vaccine to patients with cancer who have a negative SARS-CoV-2 Spike IgG at least 14 days after 2 doses of the mRNA vaccines (BNT162b2/mRNA-1273) or 28 days after the adenoviral based Ad26CoV2.S vaccine.

SUMMARY:
The goal of this study is to assess the safety and effectiveness of COVID vaccine booster doses in patients with cancer who have not developed an antibody after the U.S. Food and Drug Administration (FDA) Emergency Use Authorized COVID primary vaccination series.

DETAILED DESCRIPTION:
Cancer patients show increased morbidity with COVID-19 and need effective immunization strategies. Many healthcare regulatory agencies recommend administering 'booster' doses of COVID-19 vaccines beyond the standard two-dose series, for this group of patients. Therefore, studying the efficacy of these additional vaccine doses against SARS-CoV-2 and variants of concern is of utmost importance in this immunocompromised patient population.

The investigator team designed a prospective single arm clinical trial for consenting patients with cancer who had received two doses of mRNA, or one dose of AD26.CoV2.S vaccine, and were administered a third dose of mRNA vaccine. Patients who had no or low responses to three mRNA COVID vaccines were administered a fourth dose of mRNA vaccine. Efficacy was assessed by changes in anti-spike antibody, T-cell activity, and neutralization activity, at baseline and 4 weeks.

First Booster Dose ("3rd dose") study:

Following the informed consent process patients are enrolled into the study. After drawing baseline laboratory samples that include spike antibody, a sample for T-cell assay, and a biobank sample, patients will receive a third mRNA vaccine (initially BNT162b2 per protocol, later amended to allow for a third mRNA-1273 vaccine after the Food and Drug Administration [FDA] authorized 'booster' doses in the fall of 2021). Patients who had received Ad26.CoV2.S vaccine will receive a BNT162b2 booster vaccine. Follow-up visits are scheduled at ~4 weeks and 4-6 months following the booster dose and laboratory sample collections will be repeated.

Second Booster Dose ("4th dose") study:

For patients who did not seroconvert after three doses or had low antibody response (<1000 AU/mL as determined by in-house Abbott assay), it was hypothesized that a 'mix and match' strategy with a 2nd booster dose ("4th dose") of COVID-19 vaccine would induce seroconversion and improve boosting of humoral antibody responses. To study this, a protocol was designed wherein patients who had received their 1st booster dose ("3rd dose") of mRNA vaccines and had undetectable anti-S antibody or had an anti-S antibody level of <1000 AU/mL measured at least 14 days after third dose would be randomized to an mRNA vs. adenoviral booster ("4th") vaccine dose. Responses would be then assessed at 4 weeks after the 2nd booster dose ("4th dose") through measurement of anti-S antibody results. Complete blood counts (CBC), quantitative immunoglobulin levels (IgG, IgA, and IgM), lymphocyte subsets, T-cell responses, and neutralization activity at baseline and 4 weeks will be assessed for each of these patients. Following the implementation of this protocol, the Centers for Disease Control (CDC) published a statement that advised that the mRNA vaccines should be preferentially administered over the adenoviral vaccines given concern over rare side effects such as thrombocytopenia and thrombosis syndrome. Given this advisory, the protocol was amended to allow recruitment in a cohort that would receive a fourth dose of the BNT162b2 vaccine to comply with CDC guidelines.

ELIGIBILITY:
Inclusion Criteria (Cohort 1):

* Above the age of 18
* Meet one of the sub-criteria below:

  * Meet the CDC definition for immunocompromised status for cancer patients, i.e patients receiving active treatment for solid tumor or hematologic malignancy OR
  * Be a recipient of stem cell transplant or CAR-T cell therapy in the last 2 years OR
  * Have a negative SARS-CoV-2 spike IgG despite standard vaccination series, irrespective of active/inactive cancer status, on observation, or active therapy.
* Underwent an in-person encounter at a study facility during the study period
* Have received the second of the mRNA-based vaccines BNT162b2 and mRNA-1273 (Pfizer/BioNTech or Moderna, respectively) or one dose of the adenoviral Ad26CoV2.S (Johnson & Johnson) vaccine at least 28 days before the booster dose.

Exclusion Criteria (Cohort 1):

* Patients who have had a serious adverse reaction to any prior COVID-19 vaccines resulting in emergency room visit or hospitalization, had events related to myocarditis, thrombosis and thrombocytopenia syndrome or anaphylaxis to any prior dose of the COVID-19 vaccines.
* Patients who have had a documented COVID-19 infection in the 90 days prior to starting the study

Inclusion Criteria (Cohort 2):

* Above the age of 18
* Have a diagnosis of prior or active malignancy, either hematological or solid tumor
* Have a negative or low-level SARS-CoV-2 spike IgG after 14 days of booster vaccination series irrespective of active/inactive cancer status, on observation, or active therapy.
* Have received an FDA-authorized booster dose of mRNA (BNT162b2 and mRNA-1273) vaccine at least 28 days before study enrollment.

Exclusion Criteria (Cohort 2):

* Patients who have had a serious adverse reaction to any prior COVID-19 vaccines resulting in emergency room visit or hospitalization, had events related to myocarditis, thrombosis and thrombocytopenia syndrome or anaphylaxis to any prior dose of the COVID-19 vaccines.
* Patients who have had a documented COVID-19 infection in the 90 days prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2023-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Balazs Halmos, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thakkar A, Pradhan K, Duva B, Carreno JM, Sahu S, Thiruthuvanathan V, Campbell S, Gallego S, Bhagat TD, Rivera J, Choudhary G, Olea R, Sabalza M, Shapiro LC, Lee M, Quinn R, Mantzaris I, Chu E, Will B, Pirofski LA, Krammer F, Verma A, Halmos B. Study of efficacy and longevity of immune response to third and fourth doses of COVID-19 vaccines in patients with cancer: A single arm clinical trial. Elife. 2023 Mar 28;12:e83694. doi: 10.7554/eLife.83694. PMID 36975207

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 189 patients were assessed for eligibility to receive a booster COVID-19 vaccine after at least 28 days following completion of the standard COVID-19 vaccination series. Of the 189 patients, 56 patients declined to participate in the study, 2 patients did not meet eligibility criteria, and 25 participants were not enrolled due to 'Other reasons.' Accordingly, 106 patients were enrolled into the Booster Dose Trial.
Groups:
- Booster Dose: 1. 1st Booster Dose: Patients who have a negative SARS-CoV-2 spike IgG at least 14 days after 2 doses of the mRNA vaccines (BNT162b2 or mRNA-1273), or 28 days after the adenoviral based Ad26CoV2.S vaccine, received a third/booster mRNA vaccine (initially BNT162b2 per protocol, which was later amended to allow for third mRNA-1273 vaccine after the FDA authorized 'booster' doses in the fall of 2021). Patients then returned for follow-up at 4 weeks and 5-6 months after their third/booster dose, and their labs were repeated.
  2. 2nd Booster Dose: For patients who failed to seroconvert after their third/booster dose of vaccine or had low antibody responses (<1000 AU/mL anti-S antibody as determined by assay measured at least 14 days after the third dose) a fourth dose of either mRNA or adenoviral vaccine was administered. Responses were assessed at 4 weeks after the fourth dose to assess anti-S antibody results. Following implementation of the protocol, the Centers for Disease Control and Prevention (CDC) published a statement that advised that the mRNA vaccines should be administered preferentially over the adenoviral (Ad26.CoV2.S) vaccines.
Period: 1st Booster: 4 Week Follow up Visit
Arm/Group | Booster Dose
Started | 106
Completed | 106
Not Completed | 0
Period: 1st Booster: 4-6 Month Follow up Visit
Arm/Group | Booster Dose
Started | 106
Completed | 47
Not Completed | 59
Not completed — Lost to Follow-up | 59
Period: 2nd Booster: 4 Week Follow up Visit
Arm/Group | Booster Dose
Started (Twenty participants received a second booster dose but only 18 were enrolled. As demonstrated in the table, two patients who had received the second booster dose declined to participate.) | 20
Completed | 18
Not Completed | 2
Not completed — Declined to Participate | 2
Period: 2nd Booster: 4-6 Month Follow up Visit
Arm/Group | Booster Dose
Started | 18
Completed (Due to lack of patient participation and lack of funding the study was terminated prior to any Cohort 2 patients having reached the 4-6 month collection timepoint) | 0
Not Completed | 18

BASELINE CHARACTERISTICS:
Population: 106 participants were enrolled into the study.
Groups:
- All Study Participants: Patients who have a negative SARS-CoV-2 spike IgG at least 14 days after 2 doses of the mRNA vaccines (BNT162b2 or mRNA-1273), or 28 days after the adenoviral based Ad26CoV2.S vaccine, received a third/booster mRNA vaccine (initially BNT162b2 per protocol, which was later amended to allow for third mRNA-1273 vaccine after the FDA authorized 'booster' doses in the fall of 2021). Patients then returned for follow-up at 4 weeks and 4-6 months after their third/booster dose
Arm/Group | All Study Participants
Number analyzed (Participants) | 106
Age, Continuous [Median (Full Range); unit: years] | 68 [63.25 to 76.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 36
  African-American | 33
  Hispanic | 27
  Asian | 9
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 106
Previous Vaccine Administered [Count of Participants; unit: Participants]
  BNT162b2 | 72
  mRNA-1273 | 28
  Ad26.CoV2.S | 6
Type of Booster Vaccine [Count of Participants; unit: Participants]
  BNT162b2 | 78
  mRNA-1273 | 28
Malignancy Category [Count of Participants; unit: Participants]
  Hematologic Malignancy | 66
  Solid Tumor Malignancy | 40
Hematologic Malignancy [Count of Participants; unit: Participants] — 40 patients had solid tumors.
  Participants
    Lymphoid | 55
    Myeloid | 11
Cancer Status [Count of Participants; unit: Participants]
  Active | 69
  Progressive | 3
  Recurrent | 3
  Relapse | 7
  Remission | 24
On Treatment at the Time of Booster [Count of Participants; unit: Participants]
  Yes | 80
  No | 26
Median Titer after Primary Vaccination Series [Median (Inter-Quartile Range); unit: AU/mL] — The median titer at baseline after primary vaccination series
  AU/mL | 212.1 [50 to 2873]
Positive Anti-spike IgG Titers among Patients with evaluable T-cell Results [Count of Participants; unit: Participants] — The number of patients with evaluable T-cell immune responses at baseline was determined through a SARS-CoV-2 interferon-gamma release assay (IGRA). Population: At baseline (i.e. after primary vaccination) 88 patients had evaluable T-cell results
  Participants
    number analyzed (Participants) | 88
    (all) | 65
Patients with evaluable positive T-cell immune responses who were seronegative for Anti-S antibody [Count of Participants; unit: Participants] — Population: 65 patients with evaluable T-cell immune responses demonstrated a positive T-cell response against SARS-CoV-2
  Participants
    number analyzed (Participants) | 65
    (all) | 21
Percentage of Patients Seropositive/Seronegative at Baseline (before 1st booster dose) [Count of Participants; unit: Participants] — Population: Percentage of patients seronegative at baseline following the standard 2 dose vaccination series as demonstrated by anti-S antibody testing. Biobanked samples were available for 103 patients.
  Participants
    Seropositive Patients | 68
    Seronegative Patients | 35
Patients with neutralizing antibodies (in seropositive patients) [Count of Participants; unit: Participants] — Population: 68 patients were seropositive at baseline following primary COVID-19 vaccination series. The GenScript surrogate virus neutralization assay was used to analyze samples for neutralizing antibodies.
  Participants
    number analyzed (Participants) | 68
    (all) | 47

OUTCOME MEASURES:

1. Primary Outcome: Rate of Seroconversion for SARS-CoV-2 Spike Antibody Among Patients Who Were Seronegative After Primary Series of COVID-19 Vaccinations
Description: Rate will be determined as the percentage of patients demonstrating booster-induced seroconversion, as evidenced by anti-Spike antibody testing, who were seronegative after the primary series of FDA authorized COVID-19 vaccinations.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 35 of 106 patients were seronegative after initial 2 dose vaccination series. At 4 weeks following receipt of the booster vaccine, 57% (20/35) of these patients seroconverted and had a detectable antibody response as demonstrated by anti-S antibody testing
Measure: Count of Participants; unit: Participants
Groups:
- 1st Booster Dose: Patients who have a negative SARS-CoV-2 spike IgG at least 14 days after 2 doses of the mRNA vaccines (BNT162b2 or mRNA-1273), or 28 days after the adenoviral based Ad26CoV2.S vaccine, received a third/booster mRNA vaccine (initially BNT162b2 per protocol, which was later amended to allow for third mRNA-1273 vaccine after the FDA authorized 'booster' doses in the fall of 2021). Patients then returned for follow-up at 4 weeks and 5-6 months after their third/booster dose, and their labs were repeated.
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 35
Participants | 20

2. Primary Outcome: Percentage of Patients Who Were 'Responders' After 2nd Booster Dose
Description: A patient was classified as a responder if they either (1) had positive anti-S antibody at 4 weeks if seronegative at baseline (following 1st booster dose) or (2) if they achieved a titer of >1000 AU/mL at 4 weeks if they were sero-low at baseline (following 1st booster dose)
Time Frame: 4 weeks after administration of 2nd booster dose
Population: 18 participants were enrolled into the 2nd booster dose cohort. All 18 patients in this cohort had hematologic malignancies. 15 patients received BNT162b2 as their 2nd booster vaccine and 3 patients received Ad26.CoV2.S as their 2nd booster vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- 1st Booster Dose: For patients who failed to seroconvert after their third/booster dose of vaccine or had low antibody responses (<1000 AU/mL anti-S antibody as determined by assay measured at least 14 days after the third dose) a fourth dose of either mRNA or adenoviral vaccine was administered. Responses were assessed at 4 weeks after the fourth dose to assess anti-S antibody results. Following implementation of the protocol, the Centers for Disease Control and Prevention (CDC) published a statement that advised that the mRNA vaccines should be administered preferentially over the adenoviral (Ad26.CoV2.S) vaccines.
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 18
Participants | 12

3. Secondary Outcome: Positive Anti-Spike Antibody (IgG) Titer
Description: The number of patients with evaluable T-cell immune responses who demonstrated positive anti-S antibody (IgG) titers against SARS-CoV-2 after 1st booster dose of vaccine.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 89 patients had evaluable T-cell results at 4 weeks following 1st booster dose of vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 89
Participants | 76

4. Secondary Outcome: Spike Antibody Titer
Description: The median SARS-CoV-2 spike antibody (IgG) titer among the entire cohort at 4 weeks after administration of the 1st booster dose of vaccine was determined.
Time Frame: 4 weeks after administration of 1st booster dose
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 106
AU/mL | 9997 [880.7 to 47063]

5. Secondary Outcome: Change in Anti-Spike Antibody Titer for Patients With Hematologic Malignancies
Description: The median change in anti-S antibody titer for patients with Hematologic malignancies was determined.
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 66 patients had Hematologic malignancies
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 66
AU/mL | 2167 [0 to 10131]

6. Secondary Outcome: Change in Anti-Spike Antibody Titer for Patients With Solid Tumor Malignancies
Description: The median change in anti-S antibody titer for patients with Solid tumor malignancies was determined.
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 40 patients had Solid Tumor malignancies
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 40
AU/mL | 31010 [9531 to 44464]

7. Secondary Outcome: Change in Anti-Spike Antibody Titer Among Patients With Hematologic Malignancy by Type
Description: Median change in Anti-S antibody titers was determined in patients who presented with Hematologic (either Lymphoid or Myeloid) malignancies.
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: Of patients with Hematologic malignancies, 55 patients had Lymphoid malignancies and 11 patients had Myeloid malignancies
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 66
AU/mL
  Lymphoid Malignancies: number analyzed (Participants) | 55
  Lymphoid Malignancies | 1169 [0 to 8661]
  Myeloid Malignancies: number analyzed (Participants) | 11
  Myeloid Malignancies | 9424 [4381 to 20444]

8. Secondary Outcome: Percentage of Patients Seropositive/Seronegative Following 1st Booster Dose
Description: Percentage of Patients who were either seropositive or seronegative following administration of 1st booster dose as demonstrated by anti-S antibody testing.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 4 week samples were not collected/processed from 6 patients
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 100
Participants
  Seropositive Patients | 85
  Seronegative Patients | 15

9. Secondary Outcome: Neutralizing Antibodies Detected Among Seropositive Patients
Description: The GenScript surrogate virus neutralization assay was used to analyze samples from seropositive patients to detect for the presence of neutralizing antibodies. The percentage of patients with neutralizing antibodies was determined.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 85 patients were seropositive at 4 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 85
Participants | 77

10. Secondary Outcome: Positive T-cell Response Among Patients With a Negative Anti-S Antibody
Description: Percentage of patients with a negative anti-S antibody following 1st booster dose who demonstrated a Positive T-cell response.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 15 patients had a negative anti-S antibody result at 4 weeks following booster dose administration.
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 15
Participants | 11

11. Secondary Outcome: Positive T-cell Response Among Patients With a Negative T-cell Response at Baseline
Description: Percentage of patients who demonstrated a Positive T-cell response among those who demonstrated a negative T-cell response at baseline.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 21 patients demonstrated a negative T-cell response against SARS-CoV-2 at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 21
Participants | 14

12. Secondary Outcome: Anti-spike Antibody Titers for Patients on Anti-CD20 Antibody Therapy Within 6 Months of Treatment
Description: In order to determine association of specific cancer-directed therapies with the booster effect, median change in anti-S antibody titers were assessed for patients on anti-CD20 antibody therapy within 6 months of administration of 1st booster dose.
Time Frame: Within 6 months prior to treatment to 4 weeks after administration of 1st booster dose
Population: 25 patients were on Anti-CD20 antibody therapy within 6 months of treatment
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 25
AU/mL | 0 [0 to 0]

13. Secondary Outcome: Anti-spike Antibody Titers for Patients on Anti-CD20 Antibody Therapy
Description: In order to determine association of specific cancer-directed therapies with the booster effect, median change in anti-S antibody titers were assessed for patients on anti-CD20 antibody therapy just prior to the study.
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 25 patients were on Anti-CD20 antibody therapy just prior to the study
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 25
AU/mL | 0 [0 to 910.5]

14. Secondary Outcome: Anti-spike Antibody Titers for Patients Not on Anti-CD20 Antibody Therapy
Description: In order to determine association of specific cancer-directed therapies with the booster effect, median change in anti-S antibody titers were assessed for patients not on anti-CD20 antibody therapy just prior to the study.
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 81 patients were not on Anti-CD20 antibody therapy just prior to the study
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 81
AU/mL | 12735 [2842 to 38863]

15. Secondary Outcome: Anti-spike Antibody Titers for Patients Not on Anti-CD20 Antibody Therapy Within 6 Months of Treatment
Description: In order to determine association of specific cancer-directed therapies with the booster effect, median change in anti-S antibody titers were assessed for patients not on anti-CD20 antibody therapy within 6 months of treatment
Time Frame: Within 6 months prior to treatment to 4 weeks after administration of 1st booster dose
Population: 81 patients were not on Anti-CD20 antibody therapy within 6 months prior to treatment
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 81
AU/mL | 587 [0 to 4314]

16. Secondary Outcome: Percentage of Patients Who Remained Seropositive Following 1st Booster Dose
Description: Percentage of Patients who maintained a positive anti-S antibody (seropositive) following administration of 1st booster dose as demonstrated by anti-S antibody testing.
Time Frame: ~4-6 months after administration of 1st booster dose
Population: 47 patients completed their 4-6 month follow-up visit following 1st booster dose. All 47 were seropositive at 4 weeks. 36 of these patients had hematologic malignancies and 11 of these patients had solid malignancies. Six patients had received anti-COVID monoclonal antibody therapy as per standard of care between the 4 week and 4-6 months' follow-up period. Nine patients had received a fourth dose of COVID-19 vaccine outside of the context of the study prior to the time of 4-6 months' follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 47
Participants | 47

17. Secondary Outcome: Percentage of Seronegative Patients Before 2nd Booster Dose
Description: The percentage of patients determined to be seronegative before 2nd booster dose
Time Frame: Prior to administration of 2nd booster dose, a minimum of 14-28 days following 1st booster dose, a median of approximately 5 months
Population: 18 participants were enrolled into the second booster dose cohort. All 18 patients in this cohort had hematologic malignancies. 15 patients received BNT162b2 as their 2nd booster vaccine and 3 patients received Ad26.CoV2.S as their 2nd booster vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- 2nd Booster Dose: For patients who failed to seroconvert after their third/booster dose of vaccine or had low antibody responses (<1000 AU/mL anti-S antibody as determined by assay measured at least 14 days after the third dose) a fourth dose of either mRNA or adenoviral vaccine was administered. Responses were assessed at 4 weeks after the fourth dose to assess anti-S antibody results. Following implementation of the protocol, the Centers for Disease Control and Prevention (CDC) published a statement that advised that the mRNA vaccines should be administered preferentially over the adenoviral (Ad26.CoV2.S) vaccines.
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants | 7

18. Secondary Outcome: Percentage of Patients With Low (Anti-S Antibody) Serum Antibodies
Description: The percentage of patients with low serum antibodies before administration of the 2nd booster dose was determined by assay. Patients with anti-S antibody titers of <1000 AU/mL were determined to have low serum antibodies.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants | 11

19. Secondary Outcome: Anti-spike IgG Responders After the 2nd Booster Dose
Description: The percentage of patients who were classified as 'responders' after the 2nd Booster dose. A patient was classified as a responder if they: (1) had positive anti-S antibody at 4 weeks if seronegative after 1st booster dose or (2) if they achieved a titer of >1000 AU/mL at 4 weeks if they were sero-low after 1st booster dose.
Time Frame: ~4 weeks after administration of 2nd booster dose, a minimum of 4-6 weeks following 1st booster dose, a median of approximately 6.0-6.5 months
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants | 12

20. Secondary Outcome: Rate of Seroconversion for SARS-CoV-2 Spike Antibody Among Patients Who Remained Seronegative Following 1st Booster Dose
Description: Rate was determined as the percentage of patients demonstrating booster-induced seroconversion to positive anti-S antibody who had remained seronegative following administration of Primary Vaccination series and 1st Booster dose of BNT162b2, mRNA-1273, or AdCoV2.S COVID vaccine.
Time Frame: as for outcome 19
Population: 7 patients remained seronegative following administration of Primary vaccination series and 1st booster dose
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 7
Participants | 2

21. Secondary Outcome: Percentage of Patients With Low Anti-Spike Antibody Who Responded Following 2nd Booster Dose
Description: The percentage of Patients with low anti-Spike antibody, determined to be IgG <1000 AU/mL by assay, who responded following administration of 2nd booster dose. Responses in this context were determined to be those patients with assay results of IgG > 1000 AU/mL.
Time Frame: as for outcome 19
Population: 11 patients were sero-low (IgG <1000 AU/mL) prior to administration of 2nd booster dose
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 11
Participants | 11

22. Secondary Outcome: Anti-Spike Antibody Titer Following Administration of 1st Booster Dose
Description: The median Anti-S antibody titer following administration of the primary vaccination series and 1st booster dose in Cohort B was determined.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
AU/mL | 131.1 [50 to 432.9]

23. Secondary Outcome: Anti-Spike Antibody Titer Following Administration of 2nd Booster Dose
Description: The median Anti-S antibody titer following administration of the 2nd booster dose (Cohort B) was determined.
Time Frame: as for outcome 19
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
AU/mL | 1700 [64.3 to 18627]

24. Secondary Outcome: Positive Anti-Spike Antibody (IgG) Titer Prior to 2nd Booster Dose
Description: The number of Cohort B patients with evaluable T-cell immune responses who demonstrated positive anti-S antibody (IgG) titers against SARS-CoV-2 following 1st booster dose and prior to 2nd booster dose of vaccine.
Time Frame: as for outcome 17
Population: 14 patients in Cohort B had evaluable T-cell responses
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 14
Participants | 11

25. Secondary Outcome: Positive Anti-Spike Antibody (IgG) Titer Following 2nd Booster Dose
Description: The percentage of Cohort B patients who demonstrated positive anti-S antibody (IgG) titers against SARS-CoV-2 following administration of 2nd booster dose of vaccine.
Time Frame: as for outcome 19
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants | 17

26. Secondary Outcome: Neutralization Against Wildtype (WT) SARS-CoV-2 Variant Prior to 2nd Booster Dose
Description: Neutralization activity against the WT variant was assessed using a neutralization activity assay. The percentage of patients with positive and negative T-cell results are reported.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants
  Positive | 12
  Negative | 6

27. Secondary Outcome: Neutralization Against Wildtype (WT) SARS-CoV-2 Variant Following 2nd Booster Dose
Description: as for outcome 26
Time Frame: as for outcome 19
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants
  Positive | 13
  Negative | 5

28. Secondary Outcome: Neutralization Against Omicron BA.1 SARS-CoV-2 Variant Prior to 2nd Booster Dose
Description: Neutralization activity against the Omicron BA.1 variant was assessed using a neutralization activity assay. The percentage of patients with positive and negative T-cell results are reported.
Time Frame: as for outcome 17
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants
  Positive | 0
  Negative | 18

29. Secondary Outcome: Neutralization Against Omicron BA.1 SARS-CoV-2 Variant Following 2nd Booster Dose
Description: as for outcome 28
Time Frame: as for outcome 19
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 2nd Booster Dose
Number analyzed (Participants) | 18
Participants
  Positive | 6
  Negative | 12

30. Post Hoc Outcome: Anti-spike Antibody Titers for Patients on Bruton's Tyrosine Kinase (BTK) Inhibitors
Description: In order to determine association of specific cancer-directed therapies with the booster effect, median change in anti-S antibody titers were determined for patients on BTK inhibitors prior to the study
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 12 patients were on BTK inhibitors prior to the study
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 12
AU/mL | 0 [0 to 3393]

31. Post Hoc Outcome: Anti-spike Antibody Titers for Patients Not on Bruton's Tyrosine Kinase (BTK) Inhibitors
Description: In order to determine association of specific cancer-directed therapies with the booster effect, median change in anti-S antibody titers were determined for patients not on BTK inhibitors prior to the study
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 94 patients were not on BTK inhibitors prior to the study
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 94
AU/mL | 9355 [877.3 to 34410]

32. Post Hoc Outcome: Change in Anti-Spike Antibody Titer by Prior SARS-CoV-2 (COVID-19) Infection Status
Description: Median change in anti-S antibody titer was determined based on previous SARS-CoV-2 (COVID-19) infection status
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 9 patients had prior COVID-19 infection, 96 patients did not have prior COVID-19 infection. Prior COVID-19 infection status was unknown for 1 patient.
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 105
AU/mL
  Previous COVID-19 infection: number analyzed (Participants) | 9
  Previous COVID-19 infection | 19350 [9286 to 32151]
  No Previous COVID-19 infection: number analyzed (Participants) | 96
  No Previous COVID-19 infection | 6706 [444.1 to 33831]

33. Post Hoc Outcome: Change in Anti-Spike Antibody Titer Based on Type of Booster Administered
Description: Median change in anti-S antibody titer was determined based on the type of booster administered (BNT162b2 or mRNA-1273)
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 78 patients were administered the BNT162b2 booster and 28 patients were administered the mRNA-1273 booster
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 106
AU/mL
  BNT162b2: number analyzed (Participants) | 78
  BNT162b2 | 5534 [433.8 to 18074]
  mRNA-1273: number analyzed (Participants) | 28
  mRNA-1273 | 31451 [515.5 to 45057]

34. Post Hoc Outcome: Change in Anti-Spike Antibody Titer by Age
Description: To investigate the association of age, median change in anti-S antibody titers were determined for the cohort of patients <65 years old as opposed to the cohort of patients >=65 years old.
Time Frame: Baseline to 4 weeks after administration of 1st booster dose
Population: 106 total patients analyzed. Breakdowns by age categories described with corresponding median antibody titer results.
Measure: Median (Inter-Quartile Range); unit: AU/mL
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 106
AU/mL
  <65 years old: number analyzed (Participants) | 33
  <65 years old | 27451 [2641 to 50000]
  >=65 years old: number analyzed (Participants) | 73
  >=65 years old | 6152 [558.9 to 41765]

35. Post Hoc Outcome: Neutralization Against Wildtype (WT) SARS-CoV-2 Variant
Description: Neutralization activity against the WT variant was assessed in the seronegative cohort using a neutralization activity assay. The percentage of patients with positive and negative results are reported.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 35 patients were found be seronegative after the 1st booster dose
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 35
Participants
  Positive | 16
  Negative | 19

36. Post Hoc Outcome: Neutralization in Seronegative Cohort Against Omicron BA.1 Variant
Description: Neutralization activity against the BA.1.1529 (Omicron BA.1) variant was assessed in the seronegative cohort using a neutralization activity assay. The percentage of patients with positive and negative results are reported.
Time Frame: 4 weeks after administration of 1st booster dose
Population: 35 patients were found be seronegative after the 1st booster dose
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 35
Participants
  Positive | 6
  Negative | 29

37. Post Hoc Outcome: Percentage of Patients With Breakthrough SARS-CoV-2 Infections
Description: The percentage of patients with breakthrough SARS-CoV-2 infections was determined.
Time Frame: ~4-6 months after administration of 1st booster dose
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 47
Participants | 4

38. Post Hoc Outcome: Percentage of Patients Who Seroreverted
Description: The percentage of patients who seroreverted (i.e., no longer had detectable serum antibody) was determined
Time Frame: ~4-6 months after administration of 1st booster dose
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | 1st Booster Dose
Number analyzed (Participants) | 47
Participants | 0

ADVERSE EVENTS:
Time Frame: Through study termination, up to 6 months. Patients were observed for a minimum of 15 minutes after their booster vaccinations to monitor for adverse events. Adverse event monitoring continued via administration of a questionnaire at 4 weeks (28 days), 3 months (90 days) and 6 months (180 days) following initial booster dose administration. Additional monitoring timepoints (i.e., 12 months (365 days), and 24 months (730 days)) were not reached as the study was terminated early.
Arm/Group | Booster Dose
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 1/106
Other Adverse Events (participants affected / at risk) | 63/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Booster Dose (N=106)
Fever (General disorders) | 1 (1) — Verbatim Term: Persistent Fever. Hospitalized 3 days after booster. Listeria bacteremia unrelated to booster
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Booster Dose (N=106)
Vaccination Complication (Injury, poisoning and procedural complications) | 55 — Verbatim Terms: Sore Arm, Muscle Aches
Vaccination Site Lymphadenopathy (General disorders) | 3
Injection Site Reaction (General disorders) | 5
Nausea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 6
Fatigue (General disorders) | 9
Fever (General disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Chills (General disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 — Verbatim Term: Lower Back Pain
Dizziness (Nervous system disorders) | 3
Non-cardiac Chest Pain (General disorders) | 2 — Verbatim Term: Chest Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/22/NCT05016622/Prot_SAP_000.pdf